CLINICAL TRIAL: NCT03932331
Title: A Phase 1/2 Open Label, Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics and Clinical Efficacy of Acalabrutinib in Chinese Adult Subjects With Relapsed or Refractory Mantle Cell Lymphoma, Chronic Lymphocytic Leukemia or Other B-cell Malignancies
Brief Title: Study of Acalabrutinib in Chinese Adult Subjects With Relapsed or Refractory Mantle Cell Lymphoma, Chronic Lymphocytic Leukemia or Other B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00007; 2018L02939 (Registry Identifier: CFDA/ NMPA)
Record Dates: First submitted 2019-04-16; First posted 2019-04-30 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Phase I: Relapsed or Refractory B-cell Malignancies; Phase II Cohort A: Relapsed or Refractory Mantle Cell Lymphoma; Phase II Cohort B: Relapsed or Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib (Experimental): Acalabrutinib will be orally administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib 100 mg orally twice daily

SUMMARY:
This is an open-label, two-part study to assess the safety, tolerability, pharmacokinetics and clinical efficacy of acalabrutinib in Chinese adult subjects with R/R MCL, CLL and other B-cell malignancies. The study is divided into 2 parts: Phase 1 portion and Phase 2 portion.

ELIGIBILITY:
Inclusion Criteria

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Chinese subjects at least 18 years of age at the time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
4. Adequate hematological and organ function.
5. Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy.
6. Pathologically confirmed MCL, with documentation of chromosome translocation t(11;14) (q13;q32) and/or overexpression of cyclin D1 in association with other relevant markers (eg, CD5, CD19, CD20, PAX5). Disease had relapsed after or been refractory to previous treatment.
7. Diagnosis of CLL that meets published diagnostic criteria. Must have received ≥ 1 prior systemic therapies for CLL.
8. Active disease per iwCLL 2018 criteria that requires treatment. (CLL only)
9. Other relapsed/refractory B-cell malignancies without stand of care (phase 1 only).

Exclusion criteria

1. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject had been disease free for ≥2 years or which would not have limited survival to <2 years.
2. Significant cardiovascular disease.
3. Known central nervous system involvement of lymphoma/leukemia or leptomeningeal disease.
4. Known history of HIV, serologic status reflecting active hepatitis B or C infection.
5. Major surgery within 4 weeks before first dose of study drugs.
6. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
7. Required or received anticoagulation with warfarin or equivalent vitamin K antagonist (eg, phenprocoumon).
8. Prior exposure to a BCR or BCL-2 inhibitor.
9. Use of a strong inhibitor or inducer of CYP3A.
10. Breastfeeding or pregnant.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2026-06-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Prof, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (19):
- China (19):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Xining
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Yang S, Huang H, Zhou K, Zhao X, Han Y, Li L, Wang Y, Liu X, Li J. Acalabrutinib in Chinese patients with relapsed/refractory chronic lymphocytic leukemia: Primary analysis from an open-label, multicenter phase 1/2 trial. Ann Hematol. 2025 Jan;104(1):701-712. doi: 10.1007/s00277-024-05978-4. Epub 2024 Sep 14. PMID 39271521
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220C00007&attachmentIdentifier=8f2ee702-fd3f-49d4-b380-656845d08698&fileName=D8220c00007_CSP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220C00007&attachmentIdentifier=5ad1951f-4b52-4345-865c-b02b5439cd77&fileName=d8220c00007_CSR_Synopsis.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220C00007&attachmentIdentifier=011c5794-43d3-4a58-a570-44eb5c1dfb2c&fileName=d8220c00007_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I/II open-label study was conducted in participants with relapsed/refractory (R/R) mantle cell lymphoma (MCL), R/R chronic lymphocytic leukemia (CLL) or other B-cell malignancies at 20 study centers in China. The Phase II CLL results are reported for analysis with assessment until data cut-off (DCO) date of 18 December 2023. PD= Progressive disease.
Pre-assignment Details: This study was divided into 2 parts: Phase I portion (participants with R/R B-cell malignancies) and Phase II portion (participants with R/R MCL and R/R CLL). Study consists of screening period (28 days), treatment period until PD and a safety and survival follow-up period. A total of 105 unique participants were enrolled in the study, 12 participants in Phase I, 33 participants in Phase II MCL, 60 participants in Phase II CLL. One participant from Phase I entered Phase II MCL reporting group.
Groups:
- Phase I: Participants received single dose of acalabrutinib 100 milligram (mg) capsule orally on Day 1 Cycle 0 and followed by 2 days washout period and then received acalabrutinib 100 mg capsule orally twice daily in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Phase II MCL: Participants with MCL received acalabrutinib 100 mg capsule orally twice daily in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Phase II CLL: Participants with CLL received acalabrutinib 100 mg capsule orally twice daily in 28-day cycle until PD or specific treatment discontinuation criteria were met.
Period: Overall Study
Arm/Group | Phase I | Phase II MCL | Phase II CLL
Started | 12 | 33 | 60
Participants From Phase I Who Entered Phase II MCL | 0 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 12 | 33 | 60
Not completed — Death | 0 | 7 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Meet the point of final analysis for this cohort | 8 | 23 | 0
Not completed — Progressive disease | 3 | 0 | 0
Not completed — Lung infection | 1 | 0 | 0
Not completed — Other | 0 | 0 | 58

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all participants who received at least 1 dose of acalabrutinib. A total of 105 unique participants were enrolled in the study.
Groups:
- Phase I: Participants received single dose of acalabrutinib 100 mg capsule orally on Day 1 Cycle 0 and followed by 2 days washout period and then received acalabrutinib 100 mg capsule orally twice daily in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Phase II MCL; Phase II CLL: Participants received acalabrutinib 100 mg capsule orally twice daily in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II MCL | Phase II CLL | Total
Number analyzed (Participants) | 12 | 33 | 60 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 22 | 37 | 66
  >=65 years | 5 | 11 | 23 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 19 | 30
  Male | 5 | 29 | 41 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12 | 33 | 60 | 105

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. A SAE is an AE occurring during any study phase, that fulfils 1 or more of the following criteria: death, life-threatening, in-participant hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital abnormality or birth defect, and an important medical event that may jeopardize the participant or may require medical treatment to prevent 1 of the outcomes listed above. AEs leading to discontinuation of acalabrutinib were those with action taken was 'Drug Permanently Discontinued' for acalabrutinib.
Time Frame: From the first dose administration up to 30 days following the date of last dose of study treatment, approximately 25 months.
Population: The Safety analysis set included all participants who received at least 1 dose of acalabrutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I
Number analyzed (Participants) | 12
Participants
  Any AE | 12
  Any SAE | 2
  Any AE leading to discontinuation of Acalabrutinib | 1
  Any AE with outcome death | 0

2. Primary Outcome: Phase I: Area Under the Plasma Concentration-Time Curve From Zero to Infinity (AUCinf) of Acalabrutinib and ACP-5862 Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the AUCinf of acalabrutinib and ACP-5862 in plasma. The AUCinf was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 0 Day 1
Population: The Pharmacokinetics (PK) analysis set included all participants who received at least 1 dose of acalabrutinib with reportable acalabrutinib plasma concentration and PK parameter data with no important protocol deviations that may impact PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Phase I
Number analyzed (Participants) | 12
hour*nanogram per milliliter (h*ng/mL)
  Acalabrutinib | 1351 (47.99)
  ACP-5862 | 2421 (29.46)

3. Primary Outcome: Phase I: Area Under the Plasma Concentration-Time Curve From Zero to 12 Hours (AUC0-12) of Acalabrutinib and ACP-5862 Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the AUC0-12 of acalabrutinib and ACP-5862 in plasma. The AUC0-12 was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8 and 12 hours postdose on Cycle 0 Day 1
Population: The PK analysis set included all participants who received at least 1 dose of acalabrutinib with reportable acalabrutinib plasma concentration and PK parameter data with no important protocol deviations that may impact PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase I
Number analyzed (Participants) | 12
h*ng/mL
  Acalabrutinib | 1310 (50.39)
  ACP-5862 | 2008 (37.76)

4. Primary Outcome: Phase I: Area Under the Plasma Concentration-Time Curve From Zero to the Time of the Last Quantifiable Concentration (AUClast) of Acalabrutinib and ACP-5862 Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the AUClast of acalabrutinib and ACP-5862 in plasma. The AUClast was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 0 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase I
Number analyzed (Participants) | 12
h*ng/mL
  Acalabrutinib | 1343 (48.40)
  ACP-5862 | 2270 (32.82)

5. Primary Outcome: Phase I: Maximum Observed Plasma Drug Concentration (Cmax) of Acalabrutinib and ACP-5862 Post Single and Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the Cmax of acalabrutinib and ACP-5862 in plasma. The Cmax was determined using non-compartmental method.
Time Frame: Single dose: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8 and 12 hours postdose on Cycle 0 Day 1; Multiple dose: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I
Number analyzed (Participants) | 12
ng/mL
  Post single dose: Acalabrutinib | 967.6 (59.52)
  Post single dose: ACP-5862 | 628.1 (46.38)
  Post multiple dose: Acalabrutinib: number analyzed (Participants) | 11
  Post multiple dose: Acalabrutinib | 958.2 (60.99)
  Post multiple dose: ACP-5862 | 710.0 (38.08)

6. Primary Outcome: Phase I: Time to Reach Maximum Observed Concentration (Tmax) of Acalabrutinib and ACP-5862 Post Single and Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the tmax of acalabrutinib and ACP-5862 in plasma. The tmax was determined using non-compartmental method.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Phase I
Number analyzed (Participants) | 12
hour
  Post single dose: Acalabrutinib | 0.50 [0.48 to 1.02]
  Post single dose: ACP-5862 | 0.88 [0.73 to 2.00]
  Post multiple dose: Acalabrutinib: number analyzed (Participants) | 11
  Post multiple dose: Acalabrutinib | 0.50 [0.27 to 2.03]
  Post multiple dose: ACP-5862 | 1.00 [0.73 to 3.95]

7. Primary Outcome: Phase I: Apparent Total Body Clearance of Drug (CL/F) of Acalabrutinib Post Single and Multiple Dose of Acalabrutinib
Description: Urine samples were collected to determine the CL/F of acalabrutinib. The CL/F was determined using non-compartmental method.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Phase I
Number analyzed (Participants) | 12
liter per hour
  Post single dose | 74.01 (36.77)
  Post multiple dose | 72.81 (45.25)

8. Primary Outcome: Phase I: Apparent Volume of Distribution (Vz/F) of Acalabrutinib Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the Vz/F of acalabrutinib in plasma. The Vz/F was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 0 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Phase I
Number analyzed (Participants) | 12
liter | 171.3 (105.5)

9. Primary Outcome: Phase I: Terminal Elimination Rate Constant (λz) of Acalabrutinib and ACP-5862 Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the λz of acalabrutinib and ACP-5862 in plasma. The λz was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 0 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Phase I
Number analyzed (Participants) | 12
1/hour
  Acalabrutinib | 0.43212 (51.085)
  ACP-5862 | 0.096102 (19.036)

10. Primary Outcome: Phase I: Terminal Phase Half-Life (t1/2λz) of Acalabrutinib and ACP-5862 Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the t1/2λz of acalabrutinib and ACP-5862 in plasma. The t1/2λz was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 0 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Phase I
Number analyzed (Participants) | 12
hour
  Acalabrutinib | 1.604 (76.21)
  ACP-5862 | 7.213 (28.03)

11. Primary Outcome: Phase I: Metabolite/Parent Drug Cmax Ratio (MRCmax) of Acalabrutinib and ACP-5862 Post Single and Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the MRCmax of acalabrutinib and ACP-5862 in plasma. The MRCmax was determined using non-compartmental method.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I
Number analyzed (Participants) | 12
ratio
  Post single dose | 0.6276 (37.87)
  Post multiple dose: number analyzed (Participants) | 11
  Post multiple dose | 0.7662 (43.08)

12. Primary Outcome: Phase I: Metabolite/Parent Drug AUC Ratio (MRAUCinf) of Acalabrutinib and ACP-5862 Post Single Dose of Acalabrutinib
Description: Blood samples were collected to determine the MRAUCinf of acalabrutinib in plasma. The MRAUCinf was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 0 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I
Number analyzed (Participants) | 12
ratio | 1.732 (31.55)

13. Primary Outcome: Phase I: Area Under the Plasma Concentration-Time Curve Across the Dosing Interval (AUCτ) of Acalabrutinib and ACP-5862 Post Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the AUCτ of acalabrutinib and ACP-5862 in plasma. The AUCτ was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase I
Number analyzed (Participants) | 12
h*ng/mL
  Acalabrutinib | 1373 (43.62)
  ACP-5862 | 2707 (28.61)

14. Primary Outcome: Phase I: Minimum Observed Plasma Drug Concentration (Cmin) of Acalabrutinib and ACP-5862 Post Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the Cmin of acalabrutinib and ACP-5862 in plasma. The Cmin was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I
Number analyzed (Participants) | 12
ng/mL
  Acalabrutinib | 2.443 (148.0)
  ACP-5862 | 37.52 (37.58)

15. Primary Outcome: Phase I: Metabolite/Parent Drug AUCτ Ratio (MRAUCτ) of Acalabrutinib and ACP-5862 Post Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the MRAUCτ of acalabrutinib and ACP-5862 in plasma. The MRAUCτ was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I
Number analyzed (Participants) | 12
ratio | 1.906 (33.26)

16. Primary Outcome: Phase I: Temporal Change Parameter (TCP) in Systemic Exposure of Acalabrutinib and ACP-5862 Post Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the TCP of acalabrutinib and ACP-5862 in plasma. The TCP in systemic exposure was calculated as AUCτ (steady state)/AUCinf (first dose). The TCP was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I
Number analyzed (Participants) | 12
ratio
  Acalabrutinib | 1.017 (37.57)
  ACP-5862 | 1.118 (17.15)

17. Primary Outcome: Phase I: Accumulation Ratio of AUCτ (Rac AUC) of Acalabrutinib and ACP-5862 Post Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the Rac AUC of acalabrutinib and ACP-5862 in plasma. The Rac AUC was calculated as AUCτ (steady state)/AUCτ (first dose). The Rac AUC was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I
Number analyzed (Participants) | 12
ratio
  Acalabrutinib | 1.048 (37.97)
  ACP-5862 | 1.348 (41.64)

18. Primary Outcome: Phase I: Accumulation Ratio of Cmax (Rac Cmax) of Acalabrutinib and ACP-5862 Post Multiple Dose of Acalabrutinib
Description: Blood samples were collected to determine the Rac Cmax of acalabrutinib and ACP-5862 in plasma. The Rac Cmax was calculated as Cmax (steady state)/Cmax (first dose). The Rac Cmax was determined using non-compartmental method.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 24 and 48 hours postdose on Cycle 1 Day 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase I
Number analyzed (Participants) | 12
ratio
  Acalabrutinib: number analyzed (Participants) | 11
  Acalabrutinib | 0.8218 (59.99)
  ACP-5862 | 1.130 (70.23)

19. Primary Outcome: Phase II: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR)
Description: The ORR [based on International workshop on chronic lymphocytic leukemia (iwCLL) 2018 criteria as assessed by the BICR] was defined as the percentage of participants who achieved a complete response (CR), CR with incomplete marrow recovery (CRi), nodular partial response (nPR), and partial response (PR). The ORR and the corresponding 95% 2-sided confidence interval (CI) of ORR were presented based on Clopper-Pearson exact method.
Time Frame: Response evaluations performed at the end of Cycles 2, 4 and 6; and then every 12 weeks +/- 7 days through Cycle 25, and then every 24 weeks +/- 7 days thereafter. Assessed until 18 December 2023.
Population: Tumour response analysis set included all participants who received at least 1 dose of acalabrutinib with an available baseline tumour assessment. One participant from Phase I rolled over to Phase II MCL reporting group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 34 | 60
percentage of participants | 82.4 [65.5 to 93.2] | 86.7 [75.4 to 94.1]

20. Secondary Outcome: Phase I: Best Overall Response (BOR) Assessed by Investigator in Participants With R/R CLL
Description: The BOR is best response a participant has had following first dose date but prior to starting any subsequent anticancer therapy up to and including progression or last evaluable assessment in absence of progression. The CR: No lymph nodes >=1.5 centimeters. The CRi: Participants who fulfill all criteria for CR but have a persistent anemia, thrombocytopenia or neutropenia apparently unrelated to CLL but related to drug toxicity. The nPR: Participants who were in a complete remission but bone marrow nodules can be identified histologically. The PR: Disease >=50% from baseline. Partial response with lymphocytosis (PRL): Presence of lymphocytosis plus >=50% reduction in lymphadenopathy and/or in spleen or liver enlargement plus 1 of PR criteria for platelets or hemoglobin must be met. Stable disease (SD): Change of -49% to +49% in lymph nodes. PD: Increase >=50% from baseline or from response.
Time Frame: Response evaluations performed at the end of Cycles 2, 4 and 6; and then every 12 weeks +/- 7 days thereafter or more frequently at the investigator's discretion, approximately 25 months
Population: Tumour response analysis set included all participants who received at least 1 dose of acalabrutinib with an available baseline tumour assessment. Only participants with R/R CLL are analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I
Number analyzed (Participants) | 4
Participants
  CR | 0
  CRi | 0
  nPR | 0
  PR | 4
  PRL | 0
  SD | 0
  PD | 0
  Not evaluable | 0

21. Secondary Outcome: Phase I: Best Overall Response Assessed by Investigator in Participants With R/R MCL
Description: The BOR is best response a participant has had following first dose date but prior to starting any subsequent anticancer therapy up to and including progression or last evaluable assessment in absence of progression. CR: No lymph nodes >=1.5 centimeters. PR: Disease >=50% from baseline. SD: Change of -49% to +49% in lymph nodes. PD: Increase >=50% from baseline or from response.
Time Frame: as for outcome 20
Population: Tumour response analysis set included all participants who received at least 1 dose of acalabrutinib with an available baseline tumour assessment. Only participants with R/R MCL are analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I
Number analyzed (Participants) | 8
Participants
  CR | 1
  PR | 4
  SD | 0
  PD | 3
  Not evaluable | 0

22. Secondary Outcome: Phase II: ORR Assessed by Investigator
Description: The ORR (based on iwCLL 2018 criteria as assessed by the Investigator) was defined as the percentage of participants who achieved a CR, CRi, nPR, and PR. The ORR and the corresponding 95% 2-sided CI of ORR were presented based on Clopper-Pearson exact method.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 34 | 60
percentage of participants | 73.5 [55.6 to 87.1] | 85.0 [73.4 to 92.9]

23. Secondary Outcome: Phase II: Duration of Response (DoR) Assessed by BICR and Investigator
Description: The DoR (based on iwCLL 2018 criteria as assessed by the BICR and Investigator) was defined as the interval from the first documentation of objective response to the earlier of the first documentation of objective PD or death from any cause. The DoR was calculated using Kaplan-Meier technique.
Time Frame: as for outcome 19
Population: Tumour response analysis set included all participants who received at least 1 dose of acalabrutinib with an available baseline tumour assessment. Only participants who achieved PR or above were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 28 | 52
months
  BICR Assessment | NA [6.4 to NA] — The DOR is not mature to report median and upper limit of inter-quartile range at time of analysis. | NA [25.00 to NA] — The DOR is not mature to report median and upper limit of inter-quartile range at time of analysis.
  Investigator Assessment: number analyzed (Participants) | 25 | 51
  Investigator Assessment | NA [11.2 to NA] — The DOR is not mature to report median and upper limit of inter-quartile range at time of analysis. | NA [26.38 to NA] — The DOR is not mature to report median and upper limit of inter-quartile range at time of analysis.

24. Secondary Outcome: Phase II: Progression-Free Survival (PFS) Assessed by BICR and Investigator
Description: The PFS (based on iwCLL 2018 criteria as assessed by the BICR and Investigator) was defined as the interval from the start of acalabrutinib therapy to the earlier of the first documentation of objective PD or death from any cause. The PFS was calculated using Kaplan-Meier technique.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 34 | 60
months
  BICR Assessment | NA [5.55 to NA] — The PFS is not mature to report median and upper limit of 95% confidence interval at time of analysis. | NA [28.32 to NA] — The PFS is not mature to report median and upper limit of 95% confidence interval at time of analysis.
  Investigator Assessment | NA [5.55 to NA] — The PFS is not mature to report median and upper limit of 95% confidence interval at time of analysis. | NA [30.62 to NA] — The PFS is not mature to report median and upper limit of 95% confidence interval at time of analysis.

25. Secondary Outcome: Phase II: Time to Response (TTR) Assessed by BICR and Investigator
Description: The TTR (based on iwCLL 2018 criteria as assessed by the BICR and Investigator) was defined as the interval between the date of first dose and the date of initial documentation of a response.
Time Frame: as for outcome 19
Population: Tumour response analysis set included all participants who received at least 1 dose of acalabrutinib with an available baseline tumour assessment. Only participants with response were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 28 | 52
months
  BICR Assessment | 1.8 [1.6 to 3.7] | 5.06 [2.7 to 16.6]
  Investigator Assessment: number analyzed (Participants) | 25 | 51
  Investigator Assessment | 1.9 [1.6 to 3.7] | 5.52 [2.7 to 22.2]

26. Secondary Outcome: Phase II CLL Only: Time to Next Treatment (TTNT)
Description: The TTNT was defined as the interval from the start of acalabrutinib therapy to institution of non-protocol specified anticancer treatment for CLL or death due to any cause, whichever came first. The TTNT was calculated using Kaplan-Meier technique.
Time Frame: Response evaluations performed every 12 weeks +/- 7 days through Cycle 25, and then every 24 weeks +/- 7 days thereafter. Assessed until 18 December 2023.
Population: Tumour response analysis set included all participants who received at least 1 dose of acalabrutinib with an available baseline tumour assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II CLL
Number analyzed (Participants) | 60
months | NA [NA to NA] — The TTNT is not mature to report median and 95% confidence interval at time of analysis.

27. Secondary Outcome: Phase II CLL Only: Percentage of Participants With Minimal Residual Disease (MRD) Negativity
Description: The MRD negative rate was defined as the percentage of participants with MRD-negativity (<1 CLL cell per 10000 leukocytes) measured in the peripheral blood by flow cytometry.
Time Frame: At screening (-28 days) and end of treatment visit. Assessed until 18 December 2023.
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Phase II CLL
Number analyzed (Participants) | 60
percentage of participants | 0

28. Secondary Outcome: Phase II: Percentage of Participants With Overall Survival (OS) at Month 6
Description: The OS was defined as the interval from the start of acalabrutinib therapy to death from any cause. The OS was calculated using Kaplan-Meier technique.
Time Frame: From the first dose administration up to Month 6
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 34 | 60
percentage of participants | NA [NA to NA] — The OS is not mature to report median and 95% confidence interval at time of analysis. | 96.7 [87.3 to 99.2]

29. Secondary Outcome: Phase II: Plasma Concentration of Acalabrutinib
Description: Blood samples were collected to determine the plasma concentration of acalabrutinib.
Time Frame: At 1, 2 and 4 hours post-dose on Day 8, 15 and 22 of Cycle 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase II MCL | Phase II CLL
Number analyzed (Participants) | 33 | 60
nanogram per milliliter
  Cycle 1 Day 8: 1 hour: number analyzed (Participants) | 32 | 60
  Cycle 1 Day 8: 1 hour | 157.3 (103.6) | 238.7 (288.2)
  Cycle 1 Day 8: 2 hour | 155.0 (70.33) | 187.2 (111.4)
  Cycle 1 Day 8: 4 hour | 77.06 (94.19) | 58.73 (115.4)
  Cycle 1 Day 15: 1 hour: number analyzed (Participants) | 27 | 57
  Cycle 1 Day 15: 1 hour | 160.3 (90.00) | 206.6 (354.3)
  Cycle 1 Day 15: 2 hour: number analyzed (Participants) | 27 | 57
  Cycle 1 Day 15: 2 hour | 178.9 (70.41) | 195.7 (152.2)
  Cycle 1 Day 15: 4 hour: number analyzed (Participants) | 27 | 57
  Cycle 1 Day 15: 4 hour | 61.31 (75.60) | 49.96 (162.4)
  Cycle 1 Day 22: 1 hour: number analyzed (Participants) | 6 | 0
  Cycle 1 Day 22: 1 hour | 196.3 (93.17) |
  Cycle 1 Day 22: 2 hour: number analyzed (Participants) | 6 | 0
  Cycle 1 Day 22: 2 hour | 121.3 (87.67) |
  Cycle 1 Day 22: 4 hour: number analyzed (Participants) | 6 | 0
  Cycle 1 Day 22: 4 hour | 100.8 (162.3) |

ADVERSE EVENTS:
Time Frame: Phase I and Phase II MCL: Treatment-emergent adverse events and all-cause mortality were reported from the first dose administration up to 30 days following the date of last dose of study treatment, approximately 25 months. Phase II CLL: Treatment-emergent adverse events and all-cause mortality were reported from the first dose administration up to 30 days following the date of last dose of study treatment, approximately 41 months. Assessed until DCO 18 December 2023.
Description: The Safety analysis set included all participants who received at least 1 dose of acalabrutinib.
  Phase I and Phase II MCL: MedDRA 24.1.
Arm/Group | Phase I | Phase II MCL | Phase II CLL
All-Cause Mortality (participants affected / at risk) | 0/12 | 7/34 | 2/60
Serious Adverse Events (participants affected / at risk) | 2/12 | 6/34 | 21/60
Other Adverse Events (participants affected / at risk) | 12/12 | 28/34 | 56/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=12) | Phase II MCL (N=34) | Phase II CLL (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 6 (6)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=12) | Phase II MCL (N=34) | Phase II CLL (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (6) | 6 (8)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 12 (17)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suspected covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (6) | 8 (9) | 11 (15)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 8 (9)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 6 (11) | 8 (10)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 7 (9) | 8 (8)
Band neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Basophil count increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Bilirubin conjugated increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 2 (3)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 6 (14) | 5 (5)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 3 (5)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 4 (4)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Blood immunoglobulin a decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood immunoglobulin g decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood immunoglobulin g increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Blood immunoglobulin m decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood immunoglobulin m increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 5 (9)
Blood magnesium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (2) | 3 (4)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 5 (7)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cd19 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cd19 lymphocytes increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Cd4 lymphocytes increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cd8 lymphocytes increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Cell marker decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Complement factor c3 decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Complement factor c4 increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram p wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram pr shortened (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram q waves (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qrs complex abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram st segment abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram st segment depression (Investigations) | 0 (0) | 0 (0) | 2 (6)
Electrocardiogram st-t change (Investigations) | 0 (0) | 0 (0) | 1 (2)
Electrocardiogram st-t segment abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram high voltage (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Globulins decreased (Investigations) | 0 (0) | 0 (0) | 4 (9)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 9 (10)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 14 (20)
Helicobacter test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis b dna increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis b core antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
High density lipoprotein decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
High density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 2 (4)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 2 (5)
Lymphocyte count decreased (Investigations) | 2 (4) | 1 (2) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 8 (9) | 6 (12)
Lymphocyte percentage increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 1 (1) | 2 (4)
Natural killer cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (8) | 7 (10) | 28 (48)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 3 (5)
Non-high-density lipoprotein cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 4 (7) | 14 (19) | 24 (33)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 4 (9)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prothrombin level increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2)
Qrs axis abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 4 (11) | 8 (8) | 14 (20)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 8 (10)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (2) | 2 (4)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 3 (3)
T-lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urinary occult blood positive (Investigations) | 2 (4) | 1 (1) | 4 (4)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 5 (7) | 3 (3) | 3 (7)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 4 (5)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 3 (4)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (5)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (7)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (6) | 5 (11) | 8 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (5) | 5 (5) | 4 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Magnesium metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (7) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 7 (16) | 10 (10)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 3 (6) | 3 (3) | 4 (6)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 2 (4) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (6)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (2) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small airways disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1) | 4 (5)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 3 (5)
Purpura (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 8 (11)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Wandering pacemaker (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otolithiasis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (5)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 3 (4)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 5 (5) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 3 (5) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 5 (7) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (5) | 8 (8)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (3) | 1 (1) | 4 (5)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 4 (6)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 16 (19)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 2 (6) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Hepatitis b reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03932331/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT03932331/SAP_001.pdf